CLINICAL TRIAL: NCT00315549
Title: Multinational, Randomized, Double Blind, Comparative Study to Evaluate the Efficacy and Safety of 5 Days Telithromycin 800 mg od Versus 10 Days Penicillin V 500 mg Tid in Adolescent and Adult Subjects Equal to or Over 13 Years With Streptococcus Pyogenes Tonsillitis/Pharyngitis
Brief Title: TELI TAD - Telithromycin in Tonsillitis in Adolescents and Adults
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pediatric development program terminated by sponsor
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6134; HMR3647B/3006
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Tonsillitis; Pharyngitis
Keywords: Tonsillitis; pharyngitis; penicillin; telithromycin; ketolides; clinical trials
MeSH Terms: conditions — Tonsillitis; Pharyngitis | interventions — telithromycin; Penicillins

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Telithromycin
Drug: Penicillin

SUMMARY:
This is a multinational, randomized (1:1), double blind, comparator-controlled, 2 parallel treatment group study in subjects equal to or over 13 years of age, with Streptococcus pyogenes tonsillitis/pharyngitis (T/P). Each subject will receive either telithromycin, 400 mg over-encapsulated tablets, 800 mg once daily for 5 days or penicillin V 250 mg over-encapsulated tablets, 500 mg three times daily for 10days. Matching placebo capsules will be dispensed to maintain the blind between the treatment groups.A positive rapid identification test for streptococcal Group A antigen will be required for all subjects at Visit 1 (Day 1) for entry into the study. Throat swab specimens for bacterial culture, identification, and antibiotic-susceptibility testing will be taken at Visits 1, 3 and 4.

ELIGIBILITY:
Inclusion Criteria:

Age equal to or over 13 years;

* For female subjects, the following conditions are to be met:
* Subject is premenarchal or surgically incapable of bearing children,

  * Subject is of childbearing potential and all of the following conditions are met:
  * Have normal menstrual flow within 1 month before study entry,

    * Have negative pregnancy test (urine pregnancy test sensitive to at least 50 mU/mL, and
    * Must agree to use an accepted method of contraception throughout the study (if sexually active);
* Clinical diagnosis of acute tonsillitis/pharyngitis caused by Streptococcus pyogenes based on:

  * A positive result from a rapid detection test for Group A streptococcal antigen and submission of a throat swab specimen for bacterial culture, identification, and antibiotic-susceptibility testing; and
  * A sore and scratchy throat and/or pain on swallowing (odynophagia) together with at least 2 of the following clinical signs:

    * Tonsil and/or pharyngeal erythema and/or exudate;
    * Cervical adenopathy;
    * Uvular edema;
    * Fever

Exclusion Criteria:

* Symptoms that collectively suggest nonstreptococcal T/P (eg, laryngitis, coryza, conjunctivitis, diarrhea, cough);
* History of positive throat culture for Streptococcus pyogenes in the absence of clinical signs and symptoms of T/P;
* Infection of the deep tissues of the upper respiratory tract (eg, epiglottitis, retropharyngeal or buccal cellulitis, or abscess of the retropharynx, tonsil, or peritonsillar area) or of the suprapharyngeal respiratory tract and its connecting structures (eg, sinusitis, otitis media, or orbital/periorbital cellulitis);
* History of rheumatic heart disease;
* Known congenital prolonged QT syndrome;
* Known or suspected uncorrected hypokalemia (≤3 mmol/L [mEq/L) or hypomagnesemia or bradycardia (<50 bpm);
* Known impaired renal function, as shown by creatinine clearance ≤25 mL/min
* Myasthenia gravis;
* History of hypersensitivity or intolerance to macrolides, penicillins, or cephalosporins;
* Previous enrollment in this study or previous treatment with telithromycin;
* Children of the investigator or subinvestigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof directly involved in the conduct of the protocol.
* Is currently being treated with systemic antibacterials or has been treated with systemic antibacterials within 14 days prior to enrollment;
* Has been treated with any investigational medication within the last 30 days;
* Has been treated with rifampicin, phenytoin, carbamazepine, or St. John's wort within the last 2 weeks.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2006-02; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To compare the bacteriologic efficacy of 5-days of telithromycin to 10-days of penicillin V insubjects at the posttherapy/test-of-cure (TOC) visit in the per protocol population.

SECONDARY OUTCOMES:
To compare the bacteriologic efficacy of 5-days of telithromycin to 10-days of penicillin V insubjects at the posttherapy/test-of-cure (TOC) visit andlate posttherapy visit (Visit 4) in the bacteriologic modified intent to treat population.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (4):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, San Isidro, Buenos Aires, Argentina
- Sanofi-Aventis, Providencia, Santiago Metropolitan, Chile
- Sanofi-Aventis, San José, Costa Rica